CLINICAL TRIAL: NCT01169532
Title: A Phase I Study of Ridaforolimus and Vorinostat in Patients With Advanced Solid Tumors or Lymphoma (IND 109130)
Brief Title: Ridaforolimus and Vorinostat in Treating Patients With Advanced Solid Tumors or Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-034; NCI-2010-01907 (Registry Identifier: CTRP (Clinical Trials Reporting System))
Record Dates: First submitted 2010-07-22; First posted 2010-07-26 (Estimated); Results first posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Lymphoma; Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: conditions — Lymphoma | interventions — ridaforolimus; Vorinostat; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (ridaforolimus and vorinostat) (Experimental): Patients receive ridaforolimus PO once daily on days 1-5 and vorinostat PO twice daily on days 1-3. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: ridaforolimus; Drug: vorinostat; Procedure: biopsy; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: ridaforolimus — Given PO
  Other Names: AP23573; deforolimus; MK8669
Drug: vorinostat — Given PO
  Other Names: L-001079038; SAHA; suberoylanilide hydroxamic acid; Zolinza
Procedure: biopsy — Optional correlative studies
  Other Names: biopsies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I trial is studying the side effects and best dose of giving ridaforolimus and vorinostat together in treating patients with advanced solid tumors or lymphoma. Giving ridaforolimus in combination with vorinostat may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine which dose combinations of Ridaforolimus and Vorinostat are safe and tolerable.

II. To define the maximum tolerated dose. III. To characterize dose limiting toxicities.

SECONDARY OBJECTIVES:

I. To describe the activity of this combination amongst all enrolled patients in terms of response rate, progression free survival and overall survival.

II. To describe the activity of this combination in the subset of patients with RCC in terms of response rate, progression free survival and overall survival.

III. To describe the pharmacodynamic effects of these agents in combination.

OUTLINE: This is a dose escalation study.

Patients receive ridaforolimus orally (PO) once daily on days 1-5 and vorinostat PO twice daily on days 1-3. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every three months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological confirmation of a solid, malignant tumor or lymphoma that is refractory to standard therapies or for which no standard therapies exist
* Patients must have received at least one prior systemic therapy
* Measureable disease by RECIST v 1.1
* ECOG PS 0 or 1
* ANC >= 1500/uL
* Hgb >= 9 g/dL
* Platelets >= 100,000/uL
* AST/SGOT and ALT/SGPT =< 2.5 x upper limit of normal (ULN) or =< 5.0 x ULN in patients with liver metastases
* Total Bilirubin =< 1.5 times ULN
* Creatinine =< 2.0 mg/dL or Creatinine Clearance (calculated or 24 hour urine) >= 50 ml/min
* Female patients of childbearing potential must have a negative serum or urine pregnancy test =< 21 days of study enrollment and agree to use an effective method of contraception for the duration of the study
* Ability to understand and willingness to sign written informed consent

Exclusion Criteria:

* Prior anti-cancer treatment with either an mTOR inhibitor (i.e. temsirolimus, everolimus), or an HDAC inhibitor (i.e. Vorinostat)
* Patients who have received bevacizumab =< 6 weeks prior to day 1 of study treatment; patients who have received other chemotherapy, immunotherapy, or radiotherapy =< 3 weeks prior to day 1 of study treatment or those who have not recovered from acute adverse events due to agents administered >= 3 weeks earlier; for patients receiving targeted therapy, treatment must be discontinued at least five half-lives prior to initiation of day 1 of study treatment
* Patients who have taken valproic acid =< 2 weeks of study enrollment; valproic acid is another HDAC inhibitor
* Patients who are pregnant, plan to become pregnant, or are breastfeeding
* History of gastrointestinal bleeding within1 month of enrollment
* Serum cholesterol >= 350 mg/dL or serum triglycerides >= 400 mg/d
* Poorly controlled Type 1 or 2 diabetes, defined as hemoglobin A1C greater than 8% or a fasting glucose of > 160 mg/dL
* Active infection requiring antibiotics
* Anaphylactic reaction to macrolide antibiotics, Tween 80 (polysorbate 80)
* Patients who are not adequately recovered from a prior surgical procedure or major surgical procedure within 2 weeks prior to the first dose of study drug
* Myocardial infarction of unstable angina within 3 months of study entry
* NY Heart Association class III or IV congestive heart failure
* Known active parenchymal brain metastases; patients who have had brain metastases resected, or have received radiation therapy ending > 4 weeks prior to study entry are eligible if they meet all of the following criteria: 1) residual neurologic symptoms < grade 1, 2) no steroid requirement, 3) a follow-up MRI shows regression or stability of lesions after treatment, with no new lesions appearing
* Unable to swallow whole pills
* A requirement for one of the prohibited medications; if patient is currently taking one of these medications, they may be eligible so long as they discontinue the prohibited medication prior to starting study treatment and remain off for the duration they are taking study treatment
* Known diagnosis of HIV
* Concurrent malignancies are excluded with the following exceptions: basal cell skin cancer is allowed; cervical carcinoma in situ is allowed; any malignancy that does not require active treatment, and from which the patient has been disease free for >= 3 years is allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-10; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Plimack, Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Rockledge, Pennsylvania, United States

REFERENCES:
- [Result] Zibelman M, Wong YN, Devarajan K, Malizzia L, Corrigan A, Olszanski AJ, Denlinger CS, Roethke SK, Tetzlaff CH, Plimack ER. Phase I study of the mTOR inhibitor ridaforolimus and the HDAC inhibitor vorinostat in advanced renal cell carcinoma and other solid tumors. Invest New Drugs. 2015 Oct;33(5):1040-7. doi: 10.1007/s10637-015-0261-3. Epub 2015 Jun 20. PMID 26091915

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Ridaforolimus and Vorinostat)
Started | 16
Completed | 15
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Ridaforolimus and Vorinostat)
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 10
Age, Continuous [Median (Full Range); unit: years] | 66 [57 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: MTD denoted as the highest dose at which no more than one of six patients experienced a dose limiting toxicity (DLT), and expanded to a total of 12 patients. Any drug-related grade 3 or 4 toxicity occurring during the first three weeks of treatment (except nausea, vomiting, diarrhea, serum lipid elevation, or transient electrolyte abnormality that resolved to a grade of 0-2 with medical management) was considered a dose limiting toxicity (DLT). Assessed by National Cancer Institute (NCI) Common Terminology for Adverse Events (CTCAE) version 4.0.
Time Frame: First 3 weeks of treatment
Measure: Number; unit: milligrams
Arm/Group | Treatment (Ridaforolimus and Vorinostat)
Number analyzed (Participants) | 15
milligrams
  Ridaforolimus qd days 1-5 every week | 20
  Vorinostat bid days 1-3 every week | 100

2. Secondary Outcome: Progression Free Survival
Description: Kaplan Meier curves will be used. Proportions, 95% confidence intervals, and cumulative incidence curves will be used to characterize response rates.
Time Frame: 1 year
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Treatment (Ridaforolimus and Vorinostat)
Number analyzed (Participants) | 15
weeks | 17.1 [6.6 to 21.4]

3. Secondary Outcome: Overall Survival
Description: as for outcome 2
Time Frame: 1 year
Population: Upper limit of confidence interval not reached because at least one patient was still alive at time of data cut-off. Upper limit given is amount of time (in weeks) of overall survival at data cut-off point.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Treatment (Ridaforolimus and Vorinostat)
Number analyzed (Participants) | 15
weeks | 40.7 [28.3 to 162]

ADVERSE EVENTS:
Time Frame: 162 weeks
Arm/Group | Treatment (Ridaforolimus and Vorinostat)
All-Cause Mortality (participants affected / at risk) | 10/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 12/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Ridaforolimus and Vorinostat) (N=15)
Oral Mucositis (Gastrointestinal disorders) | 12
Fatigue (General disorders) | 11
Anorexia (Metabolism and nutrition disorders) | 11
Thrombocytopenia (Blood and lymphatic system disorders) | 11
Hyperglycemia (Metabolism and nutrition disorders) | 9
Anemia (Blood and lymphatic system disorders) | 9
Diarrhea (Gastrointestinal disorders) | 7
Nausea (Gastrointestinal disorders) | 6
weight loss (Metabolism and nutrition disorders) | 6
Elevated AST (Investigations) | 6
hypertriglyceridemia (Metabolism and nutrition disorders) | 6
Elevated ALT (Investigations) | 5
Dysguesia (General disorders) | 5
Rash, Maculo-Papular (Skin and subcutaneous tissue disorders) | 5
Neutropenia (Blood and lymphatic system disorders) | 4
Elevated Creatinine (Investigations) | 4
Constipation (Gastrointestinal disorders) | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes